CLINICAL TRIAL: NCT03523299
Title: Pilot Study to Define the Immune Response Following Cryoablation of Invasive Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator wishes to revisit design and start a new study
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIB16134; IRB00077843 (Other: JHMIRB)
Record Dates: First submitted 2018-04-05; First posted 2018-05-14 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Invasive Ductal Carcinoma, Breast
Keywords: invasive ductal carcinoma; breast cancer; cryoablation
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Breast Neoplasms | interventions — Cryosurgery; Cryotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoablation (Experimental): Participants in this arm will receive cryoablation of their breast tumor two weeks before their routine lumpectomy. They will undergo two blood draws: one before cryoablation (at the time of consent) and one after cryoablation (at the time of surgery).
  Interventions: Procedure: Cryoablation
- Control (No Intervention): Participants in this arm will undergo a blood draw at the time of consent and then will continue with their scheduled lumpectomy (standard of care).

INTERVENTIONS:
Procedure: Cryoablation — Cryoablation is a non-surgical, minimally invasive freezing procedure used to destroy tumors. In the breast, cryoablation is performed under ultrasound guidance. Due to the analgesic properties of freezing, no IV sedation or anesthesia is required. After administration of local anesthetic, the physician makes a 2-3 mm incision and inserts needle-like cryoprobes into the tumor, commencing a number of freeze-thaw cycles. Then the probe is removed, pressure is applied to the area, and a bandage is placed. The patient leaves the office without stitches and minimal, if any, pain. Any residual pain after the procedure is routinely treated with over the counter analgesics such as acetaminophen.
  Other Names: cryosurgery; cryotherapy
  Arms: Cryoablation

SUMMARY:
This study will investigate the safety, feasibility, and immune response associated with cryoablation of early invasive breast cancer prior to lumpectomy. Based on mouse models, the investigators believe that cryoablation will initiate a stronger immune response relative to the control group.

Consenting patients will be randomized to one of two arms: standard of care (control) or cryoablation (intervention). Participants will undergo a blood draw at the time of consent. Those in the control arm will continue with their standard of care lumpectomy. The intervention arm will receive cryoablation 2 weeks before their scheduled lumpectomy and undergo a second blood draw before the lumpectomy.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound visible invasive ductal carcinoma (IDC) diagnosed by core needle biopsy;
* Tumor visible by ultrasound at time of treatment;
* Unifocal primary disease;
* Tumor size between 0.5 cm and 2.0 cm (as measured on ultrasound);
* Tumor depth ≥ 0.5 cm from the skin or nipple-areola complex;
* Planned lumpectomy

Exclusion Criteria:

* Pregnant patients
* Multifocal or metastatic disease
* Planned neoadjuvant chemotherapy or radiation
* Extensive ductal carcinoma in situ (DCIS; >25% DCIS component) either diagnosed on core biopsy or strongly suggested by imaging
* Known allergy to both lidocaine and benzocaine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events [safety] | 1 day after cryoablation
  Assessed via phone call with participant and including any participant-reported adverse events, such as pain, bruising, bleeding, swelling, and skin changes
Immune response | One week after lumpectomy
  Immunohistochemical analysis of biomarkers in blood and resected tissue
Cosmetic outcome | Change from one month to one year after lumpectomy
  Change in appearance based on distortion and volume loss of the breast
Tumor margin status [effectiveness] | 7-10 days after lumpectomy
  Assessment of whether excised tumor's margins are positive or negative for cancer, and whether re-excision is required

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Santa-Maria, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT03523299/Prot_SAP_001.pdf